CLINICAL TRIAL: NCT06482203
Title: Comparison of Trunk Extensor Endurance Training Versus Scapular Mobilization in Patient With Thoracic Kyphosis.
Brief Title: Trunk Extensor Endurance Training Versus Scapular Mobilization in Patient With Thoracic Kyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/MS-PT/01678
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Thoracic Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(Trunk Extensor Endurance Training) (Experimental): Trunk Extensor Endurance Training Level 1: Prone shoulder extension or prone shoulder raises Level 2: Prone back extension Level 3: Prone Ys or Y raises Level 4:Superman pose Level 5:Superman or prone cobra (The given position should be hold for 10 seconds and performs 25 repetitions with 3 sec rests in between the efforts)
  Interventions: Other: Trunk Extensor Endurance training & Scapular mobilization
- Group 2(Scapular Mobilization) (Experimental): Patient side lying. This intervention program includes, supero-inferior, medio-lateral along with circumduction movements.
  Procedure:
  Patients were side lying with their arms in 90°flexion during scapula mobilization.
  The physiotherapist completed 3 sets of 10-15 repetitions of each of the supero-inferior, medio-lateral, and circumduction movements while holding the scapula from the medial border. Between each session, there was a 10 or 30-second break. The length of rests was adjusted depending on the patient's endurance and comfort.
  Interventions: Other: Trunk Extensor Endurance training & Scapular mobilization

INTERVENTIONS:
Other: Trunk Extensor Endurance training & Scapular mobilization — Trunk Extensor Endurance Training Level 1:Prone shoulder extension or prone shoulder raises Level 2: Prone back extension Level 3: Prone Ys or Y raises Level 4:Super man pose Level 5:Super man or prone cobra
  (The given position should be hold for 10 seconds and performs 25 repetitions with 3 sec rests in between the efforts)
  Scapular Mobilization:
  Intervention program includes, supero-inferior, medio-lateral along with circumduction movements).
  3 sets of 10-15 repetitions of each of the supero-inferior ,medio-lateral, and circumduction movements Between each session, there was a10 or 30-second break. The length of rests was adjusted depending on the patient's endurance

SUMMARY:
To compare the effect of Trunk extensor endurance training and scapular mobilization on thoracic pain in patient with thoracic kyphosis.

To compare the effect of Trunk extensor endurance training and scapular mobilization on kyphotic angle in patient with thoracic kyphosis To compare the effect of Trunk extensor endurance training and scapular mobilization on shoulder ROM in patient with thoracic kyphosis

ELIGIBILITY:
Inclusion Criteria:

* Both gender (Male and female)
* Age 20-40
* Postural kyphosis
* Kyphotic angle exceeds 40°
* Thoracic pain>3

Exclusion Criteria:

* Thoracic, Scapular and clavicle abnormalities
* Vertebral fractures, history of trauma or spinal surgery
* History of prolonged use steroid (more than 6 months),rheumatologic conditions
* Cardiac, autoimmune diseases
* Structural kyphosis(X-ray findings)
* Scoliosis(x-ray findings)
* Cancer, neurological disorders, metastasis, or inflammatory
* Osteoporosis, Pregnancy or any genetic conditions affecting their bones, muscles or cartilage.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12-07 (Estimated); Study Completion 2024-12-07 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  Thoracic pain will be measure through Numeric pain rating scale, 0 no pain 10 maximum pain
kyphotic angle | 4 weeks
  Inclinometer will be used to measure the angle
Shoulder ROM | 4 weeks
  Goniometer is used to measure the Shoulder all range of motion (ROM)

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila Yaqub, masters, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital(LRH), Peshawar, Khyber Pakhutunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng Q, Wang M, Zhang Y, Zhou Y. The effect of a corrective functional exercise program on postural thoracic kyphosis in teenagers: a randomized controlled trial. Clin Rehabil. 2018 Jan;32(1):48-56. doi: 10.1177/0269215517714591. Epub 2017 Jun 14. PMID 28610442
- [Background] Yaman O, Dalbayrak S. Kyphosis and review of the literature. Turk Neurosurg. 2014;24(4):455-65. doi: 10.5137/1019-5149.JTN.8940-13.0. PMID 25050667
- [Background] Graham P. Scheuermann's Kyphosis. Orthop Nurs. 2023 Jan-Feb 01;42(1):53-55. doi: 10.1097/NOR.0000000000000914. No abstract available. PMID 36702097
- [Background] Etemadifar MR, Mahdinezhad Yazdi M. Evaluation of changes in kyphosis angle, apex and quality of life of patients with Scheuermann kyphosis using Kyphologic brace. Int J Physiol Pathophysiol Pharmacol. 2022 Jun 15;14(3):187-192. eCollection 2022. PMID 35891934
- [Background] Sato T, Koizumi M, Kim JH, Kim JH, Wang BJ, Murakami G, Cho BH. Fetal development of deep back muscles in the human thoracic region with a focus on transversospinalis muscles and the medial branch of the spinal nerve posterior ramus. J Anat. 2011 Dec;219(6):756-65. doi: 10.1111/j.1469-7580.2011.01430.x. Epub 2011 Sep 29. PMID 21954879
- [Background] Yoo WG. Effects of thoracic posture correction exercises on scapular position. J Phys Ther Sci. 2018 Mar;30(3):411-412. doi: 10.1589/jpts.30.411. Epub 2018 Mar 2. PMID 29581661
- [Background] Park SY, Yoo WG. Effect of sustained typing work on changes in scapular position, pressure pain sensitivity and upper trapezius activity. J Occup Health. 2013;55(3):167-72. doi: 10.1539/joh.12-0254-oa. Epub 2013 Apr 13. PMID 23585498
- [Background] Park SJ, Kim SH, Kim SH. Effects of Thoracic Mobilization and Extension Exercise on Thoracic Alignment and Shoulder Function in Patients with Subacromial Impingement Syndrome: A Randomized Controlled Pilot Study. Healthcare (Basel). 2020 Sep 2;8(3):316. doi: 10.3390/healthcare8030316. PMID 32887287
- [Background] Lewis JS, Valentine RE. Clinical measurement of the thoracic kyphosis. A study of the intra-rater reliability in subjects with and without shoulder pain. BMC Musculoskelet Disord. 2010 Mar 1;11:39. doi: 10.1186/1471-2474-11-39. PMID 20193055
- [Background] Sibson BE, Tobolsky VA, Kistner TM, Holowka NB, Jemutai J, Sigei TK, Ojiambo R, Okutoyi P, Lieberman DE. Trunk muscle endurance, strength and flexibility in rural subsistence farmers and urban industrialized adults in western Kenya. Am J Hum Biol. 2022 Feb;34(2):e23611. doi: 10.1002/ajhb.23611. Epub 2021 May 14. PMID 33988283
- [Background] Ogaya S, Suzuki M, Yoshioka C, Nakamura Y, Kita S, Watanabe K. The effects of trunk endurance training on running kinematics and its variability in novice female runners. Sports Biomech. 2024 Aug;23(8):997-1008. doi: 10.1080/14763141.2021.1906938. Epub 2021 Apr 28. PMID 33906577
- [Background] Duzgun I, Turgut E, Eraslan L, Elbasan B, Oskay D, Atay OA. Which method for frozen shoulder mobilization: manual posterior capsule stretching or scapular mobilization? J Musculoskelet Neuronal Interact. 2019 Sep 1;19(3):311-316. PMID 31475938
- [Background] Zappala M, Lightbourne S, Heneghan NR. The relationship between thoracic kyphosis and age, and normative values across age groups: a systematic review of healthy adults. J Orthop Surg Res. 2021 Jul 9;16(1):447. doi: 10.1186/s13018-021-02592-2. PMID 34243795
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Moffroid MT, Haugh LD, Haig AJ, Henry SM, Pope MH. Endurance training of trunk extensor muscles. Phys Ther. 1993 Jan;73(1):10-7. PMID 8417455
- [Background] Chok B, Lee R, Latimer J, Tan SB. Endurance training of the trunk extensor muscles in people with subacute low back pain. Phys Ther. 1999 Nov;79(11):1032-42. PMID 10534796